CLINICAL TRIAL: NCT00781430
Title: An Open-Label, Single-Dose, Parallel-Group Study Of The Pharmacokinetics And Safety Of Neratinib In Subjects With Chronic Hepatic Impairment And In Matched Healthy Adults
Brief Title: Study Evaluating The PK And Safety Of Neratinib In Healthy Subjects And Subjects With Chronic Liver Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 3144A1-1111; B1891009
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Hepatic Insufficiency
MeSH Terms: conditions — Hepatic Insufficiency | interventions — neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Neratinib (HKI-272)

INTERVENTIONS:
Drug: Neratinib (HKI-272) — Neratinib 40-mg oral tablets. SINGLE DOSE of 120-mg (3 x 40-mg tablets)

SUMMARY:
The purpose of this study is to assess the pharmacokinetics of neratinib and to assess the safety and tolerability of neratinib in healthy subjects and subjects with chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of nonchildbearing potential (WONCBP) aged 18 to 65 years inclusive at screening.

WONCBP may be included if they are either surgically sterile (hysterectomy or oophorectomy) or postmenopausal for =1 year (with follicle-stimulating hormone [FSH] level =38 mIU/mL) and must have a negative serum pregnancy test result within 48 hours before administration of test article. 2-Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay. 3-Have a high probability for compliance with and completion of the study

Exclusion Criteria:

* Family history of QT prolongation, syncope, seizure, or unexplained cardiac-related death. 2-Presence or history of any disorder that may prevent the successful completion of the study. 3-History of drug abuse within 1 year before study day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of neratinib in healthy volunteers compared to hepatically impaired patients through analysis of blod samples collected after neratinib administration in these 2 populations. | 4 weeks

SECONDARY OUTCOMES:
Safety based on adverse events monitoring, physical examinations, vital sign evaluations, 12-lead ECGs and routine laboratory tests. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (1):
- Pfizer Investigational Site, Moscow, Russia